CLINICAL TRIAL: NCT03489226
Title: A Pilot Study of the Effect of a Dietary Herbal Supplement Containing Capsaicin or Placebo on Satiety, Metabolic Rate and Food Intake in Healthy Adults.
Brief Title: Capsimax Effect on Metabolic Rate, Satiety and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Medical Director and Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2016-011
Record Dates: First submitted 2017-12-18; First posted 2018-04-05 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Energy Metabolism; Eating; Hunger
Keywords: capsaicin; energy expenditure; satiety; food intake
MeSH Terms: interventions — Meals

STUDY DESIGN:
Intervention Model Description: 4 arm crossover trial
Who Masked: Participant, Investigator
Masking Description: Supplement and placebo capsules with identical appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Capsimax 2 mg (Active Comparator): single dose with satiety measures and metabolic rate measured before and after. Food intake measured 1 hour after dose.
  Interventions: Dietary Supplement: Capsimax
- Placebo (Placebo Comparator): single dose with satiety measures and metabolic rate measured before and after. Food intake measured 1 hour after dose.
  Interventions: Dietary Supplement: Placebo
- Capsimax 4 mg plus 250 kcal meal (Active Comparator): single dose with 250 kcal meal with satiety measures and metabolic rate measured before and after. Food intake measured 1 hour after dose.
  Interventions: Dietary Supplement: Capsimax; Other: Meal
- Placebo plus 250 kcal meal (Placebo Comparator): single dose with 250 kcal meal with satiety measures and metabolic rate measured before and after. Food intake measured 1 hour after dose.
  Interventions: Dietary Supplement: Placebo; Other: Meal

INTERVENTIONS:
Dietary Supplement: Capsimax — Capsimax
  Arms: Capsimax 2 mg; Capsimax 4 mg plus 250 kcal meal
Dietary Supplement: Placebo — Placebo
  Arms: Placebo; Placebo plus 250 kcal meal
Other: Meal — Meal
  Arms: Capsimax 4 mg plus 250 kcal meal; Placebo plus 250 kcal meal

SUMMARY:
Comparison of Capsimax™ 2mg and 4mg of capsicum extract vs. placebo on metabolic rate and satiety.

DETAILED DESCRIPTION:
Capsimax™ is a capsicum extract in a bead technology to avoid oral and gastric burning. Capsimax™ 2mg, Capsimax™ 4 mg and placebo was initially given as a single dose on an empty stomach with measures of metabolic rate, and satiety before and after and food intake at 1 hour after Capsimax™.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 25 and 40 kg/m2 inclusive
2. Healthy
3. If of child-bearing potential, use of effective contraception

Exclusion Criteria:

Subjects excluded will:

1. Have received an investigational product in another trial within 30 days of enrollment.
2. Have lost 10 or more pounds in the 3 months prior to randomization and maintained the weight loss.
3. Use tobacco products
4. Use a nicotine patch or gum.
5. Take regular medication other than oral contraceptives or estrogen replacement therapy.
6. Take products containing ephedra or medications known to increase metabolic rate like stimulants taken for attention deficit disorder.
7. Not eat at regular mealtimes.
8. Have a history of alcohol or drug abuse in the past year.
9. Nurse a baby or be a member of a vulnerable population including adults unable to consent, pregnant women, prisoners or minors.
10. Have a clinically significant history of diabetes, high blood pressure (>140/90), thyroid disease, heart disease, kidney disease or liver disease.
11. Have a known allergy to capsaicin caffeine, piperine or niacin.
12. Have clinically significant laboratory findings in the opinion of the investigator.
13. Score greater than 13 on the restraint scale of the 3-factor eating questionnaire.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic Rate | up to 5 hours
  Metabolic cart measurement difference before and after intervention

SECONDARY OUTCOMES:
Satiety by Visual Analog Scale (hunger, fullness, prospective food intake and satisfaction) | Baseline to 4 hours
  Difference in area under the curve from baseline of the Mean Visual Analog. Each question on the scale ranges from 0 to 100 mm. The two ends of the scale are anchored by the highest and lowest values (e.g. "the hungriest I have ever been" to "no hunger at all"). Some questions have high values on the right and others have high values on the left. Each question (hunger, fullness, prospective food intake and satisfaction) is a sub-scale. Each sub-scale is scored separately.
Food Intake | 1 hour after intervention
  Meal with unlimited portions

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No